CLINICAL TRIAL: NCT00006286
Title: Treatment for Adolescents With Depression Study (TADS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: N01 MH80008; DSIR CT
Record Dates: First submitted 2000-09-14; First posted 2000-09-15 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2005-11

CONDITIONS: Major Depressive Disorder; Depression
Keywords: Depression; Major Depressive Disorder; Fluoxetine; Prozac; SSRI; Psychotherapy; CBT; Teenagers; Adolescents; Teens
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Fluoxetine; Psychotherapy

INTERVENTIONS:
Drug: Fluoxetine
Behavioral: Psychotherapy

SUMMARY:
TADS is designed to compare the effectiveness of established treatments for teenagers suffering from major depressive disorder (MDD). The treatments are: psychotherapy ("talking therapy"); medication; and the combination of psychotherapy and medication. Altogether, 432 teenagers (both males and females) ages 12 to 17, will take part in this study at 12 sites in the United States.

The TADS design will provide answers to the following questions: What is the long-term effectiveness of medication treatment of teenagers who have major depression? What is the long-term effectiveness of a specific psychotherapy ("talking therapy) in the treatment of teenagers who have major depression? How does medication treatment compare with psychotherapy in terms of effectiveness, tolerability and teenager and family acceptance? And, What is the cost-effectiveness of medication, psychotherapy and combined treatments?

The medication being used in this study is called fluoxetine. Fluoxetine is also known as Prozac. Research has shown that medications like Prozac help depression in young persons. Fluoxetine has been approved by the FDA for use in the treatment of child and adolescent (ages 7 to 17 years) depression.

The psychotherapy or "talking therapy" being used in this study is called Cognitive Behavioral Therapy (CBT). CBT is a talking therapy that will teach both the teenager and his or her family member (e.g., parent) new skills to cope better with depression. Specific topics include education about depression and the causes of depression, setting goals, monitoring mood, increasing pleasant activities, social problem-solving, correcting negative thinking, negotiation, compromise and assertiveness. CBT sessions may also help with resolving disagreements as they affect families.

DETAILED DESCRIPTION:
TADS is a randomized controlled clinical trial that will compare the effectiveness of established treatments---cognitive-behavioral psychotherapy, medication management, and their combination---for adolescents suffering from major depressive disorder (MDD).

The experimental design consists of three treatment stages and a follow-up phase. Stage I (12 weeks) is a four-group randomized comparison of four treatments: antidepressant medication alone (Fluoxetine); psychotherapy alone (CBT); a combination of the medication and psychotherapy (Comb); and a placebo control medication condition (Pbo). Stage II (six weeks) is a treatment consolidation phase in which we ask whether longer treatment in responders and higher intensity treatment in partial responders to their Stage I treatment would be helpful. Non-responders at the end of Stage I will be referred to open community treatment, or for ethical and practical reasons in the case of non-responders to Placebo, to open treatment of their choice with one of the three active study treatments administered by the study team. Responders at the end of Stage I advance to 6 weeks of maintenance treatment in their assigned arm. Partial responders to CBT receive an additional 6 weeks of CBT in their assigned arm; partial responders to Fluoxetine may receive a higher dose for six weeks. Partial responders to the Comb treatment will receive an additional 6 weeks of CBT and may receive a higher dose of medication for six weeks. Stage III (18 weeks) is a treatment maintenance phase for those teenagers who have continued to respond well. Treatment will be continued and progress will be monitored. Stage IV (one year) is an assessment-only follow-up phase to help us understand the long-term benefits of the treatments.

The recruitment strategy is designed to enter into treatment a volunteer clinical sample of 432 teenagers, both males and females, ages 12 to 17, at ten sites. A multiple gating procedure will be used in which patients will be screened, assessed for study eligibility, and if eligible, consented before randomization to one of the four treatment groups. Patients will be selected without regard to race, gender, or ethnicity and it is expected that the sample will match patients seen in general clinical practice. Patients will be recruited from multiple sources including: mental health identified children, i.e., children already coming to a clinic; primary care identified children (pediatric and family physicians); teacher or school identified children (i.e., school refers through the parents or primary caretaker); and families who self-refer.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis DSM-IV of Major Depressive Disorder, pervasive and stable; Children's Depression Rating Scale-R total score at least 45; Ages 12-17 inclusive; Grade in school: 6-12; Full-Scale IQ at least 80; Medication-free before start of study; Outpatient; Parent (or family member) involvement

Exclusion Criteria:

* Bipolar disorder; Severe Conduct Disorder; Substance Use/Abuse/Dependence; Pervasive Developmental Disorders; Thought Disorder; Suicidality or homicidality; Concurrent treatment with psychotropic drug (stable stimulant for ADHD permitted) or psychotherapy outside study; Two previous failed SSRI trials or a failed trial of CBT for depression; Intolerance to fluoxetine; Non-English speaking patient; Pregnancy or breastfeeding; No phone in home; Lack of parent or family member)involvement.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 432
Dates: Start 1998-09; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: John March, Study Director — Duke University; Anne Marie Albano, Principal Investigator — NYU Langone Health; David Rosenberg, MD, Principal Investigator — Wayne State Univ; Charles Casat, Principal Investigator — Carolinas Medical Center-Randlolph; Graham Emslie, Principal Investigator — University of Texas Soutwestern; Christopher Kratochvil, Principal Investigator — University of Nebraska; Paul Rohde and Anne Simons, Principal Investigator — University of Oregon; John Walkup, Principal Investigator — Johns Hopkins University; Elizabeth Weller, Principal Investigator — Children's Hospital of Philadelphia; Bruce Waslick, Principal Investigator — New York State Psychiatric Inst; Mark Reinecke, Principal Investigator — Northwestern University; Elizabeth Cottingham, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Norah Feeny, PhD, Principal Investigator — Case Western Reserve University
Locations (12):
- United States (12):
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York University Medical Center, New York, New York
  - New York State Psychiatric Institute, New York, New York
  - Behavioral Health Center, Charlotte, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oregon, Eugene, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Background] Glass RM. Treatment of adolescents with major depression: contributions of a major trial. JAMA. 2004 Aug 18;292(7):861-3. doi: 10.1001/jama.292.7.861. No abstract available. PMID 15316001
- [Background] Treatment for Adolescents With Depression Study Team. Treatment for Adolescents With Depression Study (TADS): rationale, design, and methods. J Am Acad Child Adolesc Psychiatry. 2003 May;42(5):531-42. doi: 10.1097/01.CHI.0000046839.90931.0D. PMID 12707557
- [Result] March J, Silva S, Petrycki S, Curry J, Wells K, Fairbank J, Burns B, Domino M, McNulty S, Vitiello B, Severe J; Treatment for Adolescents With Depression Study (TADS) Team. Fluoxetine, cognitive-behavioral therapy, and their combination for adolescents with depression: Treatment for Adolescents With Depression Study (TADS) randomized controlled trial. JAMA. 2004 Aug 18;292(7):807-20. doi: 10.1001/jama.292.7.807. PMID 15315995
- [Result] Treatment for Adolescents with Depression Study (TADS) Team. The Treatment for Adolescents With Depression Study (TADS): demographic and clinical characteristics. J Am Acad Child Adolesc Psychiatry. 2005 Jan;44(1):28-40. doi: 10.1097/01.chi.0000145807.09027.82. PMID 15608541
- [Result] March J, Silva S, Vitiello B; TADS Team. The Treatment for Adolescents with Depression Study (TADS): methods and message at 12 weeks. J Am Acad Child Adolesc Psychiatry. 2006 Dec;45(12):1393-403. doi: 10.1097/01.chi.0000237709.35637.c0. PMID 17135984
- [Result] Emslie G, Kratochvil C, Vitiello B, Silva S, Mayes T, McNulty S, Weller E, Waslick B, Casat C, Walkup J, Pathak S, Rohde P, Posner K, March J; Columbia Suicidality Classification Group; TADS Team. Treatment for Adolescents with Depression Study (TADS): safety results. J Am Acad Child Adolesc Psychiatry. 2006 Dec;45(12):1440-55. doi: 10.1097/01.chi.0000240840.63737.1d. PMID 17135989
- [Result] Curry J, Rohde P, Simons A, Silva S, Vitiello B, Kratochvil C, Reinecke M, Feeny N, Wells K, Pathak S, Weller E, Rosenberg D, Kennard B, Robins M, Ginsburg G, March J; TADS Team. Predictors and moderators of acute outcome in the Treatment for Adolescents with Depression Study (TADS). J Am Acad Child Adolesc Psychiatry. 2006 Dec;45(12):1427-39. doi: 10.1097/01.chi.0000240838.78984.e2. PMID 17135988
- [Result] Kratochvil C, Emslie G, Silva S, McNulty S, Walkup J, Curry J, Reinecke M, Vitiello B, Rohde P, Feeny N, Casat C, Pathak S, Weller E, May D, Mayes T, Robins M, March J; TADS Team. Acute time to response in the Treatment for Adolescents with Depression Study (TADS). J Am Acad Child Adolesc Psychiatry. 2006 Dec;45(12):1412-8. doi: 10.1097/01.chi.0000237710.73755.14. PMID 17135986
- [Result] Kennard B, Silva S, Vitiello B, Curry J, Kratochvil C, Simons A, Hughes J, Feeny N, Weller E, Sweeney M, Reinecke M, Pathak S, Ginsburg G, Emslie G, March J; TADS Team. Remission and residual symptoms after short-term treatment in the Treatment of Adolescents with Depression Study (TADS). J Am Acad Child Adolesc Psychiatry. 2006 Dec;45(12):1404-11. doi: 10.1097/01.chi.0000242228.75516.21. PMID 17135985
- [Result] Vitiello B, Rohde P, Silva S, Wells K, Casat C, Waslick B, Simons A, Reinecke M, Weller E, Kratochvil C, Walkup J, Pathak S, Robins M, March J; TADS Team. Functioning and quality of life in the Treatment for Adolescents with Depression Study (TADS). J Am Acad Child Adolesc Psychiatry. 2006 Dec;45(12):1419-26. doi: 10.1097/01.chi.0000242229.52646.6e. PMID 17135987
- [Result] March JS, Silva S, Petrycki S, Curry J, Wells K, Fairbank J, Burns B, Domino M, McNulty S, Vitiello B, Severe J. The Treatment for Adolescents With Depression Study (TADS): long-term effectiveness and safety outcomes. Arch Gen Psychiatry. 2007 Oct;64(10):1132-43. doi: 10.1001/archpsyc.64.10.1132. PMID 17909125
- [Result] Herman KC, Ostrander R, Walkup JT, Silva SG, March JS. Empirically derived subtypes of adolescent depression: latent profile analysis of co-occurring symptoms in the Treatment for Adolescents with Depression Study (TADS). J Consult Clin Psychol. 2007 Oct;75(5):716-28. doi: 10.1037/0022-006X.75.5.716. PMID 17907854
- [Derived] Jureidini J, Moncrieff J, Klau J, Aboustate N, Raven M. Treatment guesses in the Treatment for Adolescents with Depression Study: Accuracy, unblinding and influence on outcomes. Aust N Z J Psychiatry. 2024 Apr;58(4):355-364. doi: 10.1177/00048674231218623. Epub 2023 Dec 21. PMID 38126083
- [Derived] Baumgartner N, Foster S, Emery S, Berger G, Walitza S, Haberling I. How Are Discrepant Parent-Child Reports Integrated? A Case of Depressed Adolescents. J Child Adolesc Psychopharmacol. 2021 May;31(4):279-287. doi: 10.1089/cap.2020.0116. Epub 2020 Dec 29. PMID 33373537
- [Derived] Wang B, Ogburn EL, Rosenblum M. Analysis of covariance in randomized trials: More precision and valid confidence intervals, without model assumptions. Biometrics. 2019 Dec;75(4):1391-1400. doi: 10.1111/biom.13062. Epub 2019 Jun 3. PMID 31009064
- [Derived] Foster S, Mohler-Kuo M, Tay L, Hothorn T, Seibold H. Estimating patient-specific treatment advantages in the 'Treatment for Adolescents with Depression Study'. J Psychiatr Res. 2019 May;112:61-70. doi: 10.1016/j.jpsychires.2019.02.021. Epub 2019 Feb 28. PMID 30856378
- [Derived] Scott K, Lewis CC, Marti CN. Trajectories of Symptom Change in the Treatment for Adolescents With Depression Study. J Am Acad Child Adolesc Psychiatry. 2019 Mar;58(3):319-328. doi: 10.1016/j.jaac.2018.07.908. Epub 2019 Jan 8. PMID 30768414
- [Derived] Foster S, Mohler-Kuo M. Treating a broader range of depressed adolescents with combined therapy. J Affect Disord. 2018 Dec 1;241:417-424. doi: 10.1016/j.jad.2018.08.027. Epub 2018 Aug 12. PMID 30145512
- [Derived] Lewis CC, Simons AD, Nguyen LJ, Murakami JL, Reid MW, Silva SG, March JS. Impact of childhood trauma on treatment outcome in the Treatment for Adolescents with Depression Study (TADS). J Am Acad Child Adolesc Psychiatry. 2010 Feb;49(2):132-40. doi: 10.1097/00004583-201002000-00007. PMID 20215935
- [Derived] Kratochvil CJ, May DE, Silva SG, Madaan V, Puumala SE, Curry JF, Walkup J, Kepley H, Vitiello B, March JS. Treatment response in depressed adolescents with and without co-morbid attention-deficit/hyperactivity disorder in the Treatment for Adolescents with Depression Study. J Child Adolesc Psychopharmacol. 2009 Oct;19(5):519-27. doi: 10.1089/cap.2008.0143. PMID 19877976
- [Derived] Treatment for Adolescents With Depression Study (TADS) Team; March J, Silva S, Curry J, Wells K, Fairbank J, Burns B, Domino M, Vitiello B, Severe J, Riedal K, Goldman M, Feeny N, Findling R, Stull S, Baab S, Weller EB, Robbins M, Weller RA, Jessani N, Waslick B, Sweeney M, Dublin R, Walkup J, Ginsburg G, Kastelic E, Koo H, Kratochvil C, May D, LaGrone R, Vaughan B, Albano AM, Hirsch GS, Podniesinki E, Chu A, Reincecke M, Leventhal B, Rogers G, Jacobs R, Pathak S, Wells J, Lavanier SA, Danielyan A, Rohde P, Simons A, Grimm J, Frank S, Emslie G, Kennard B, Hughes C, Mayes TL, Rosenberg D, Benazon N, Butkus M, Bartoi M. The Treatment for Adolescents With Depression Study (TADS): outcomes over 1 year of naturalistic follow-up. Am J Psychiatry. 2009 Oct;166(10):1141-9. doi: 10.1176/appi.ajp.2009.08111620. Epub 2009 Sep 1. PMID 19723787
- [Derived] Domino ME, Foster EM, Vitiello B, Kratochvil CJ, Burns BJ, Silva SG, Reinecke MA, March JS. Relative cost-effectiveness of treatments for adolescent depression: 36-week results from the TADS randomized trial. J Am Acad Child Adolesc Psychiatry. 2009 Jul;48(7):711-720. doi: 10.1097/CHI.0b013e3181a2b319. PMID 19465880
- [Derived] Rohde P, Silva SG, Tonev ST, Kennard BD, Vitiello B, Kratochvil CJ, Reinecke MA, Curry JF, Simons AD, March JS. Achievement and maintenance of sustained response during the Treatment for Adolescents With Depression Study continuation and maintenance therapy. Arch Gen Psychiatry. 2008 Apr;65(4):447-55. doi: 10.1001/archpsyc.65.4.447. PMID 18391133
- [Derived] Vitiello B, Kratochvil CJ, Silva S, Curry J, Reinecke M, Pathak S, Waslick B, Hughes CW, Prentice ED, May DE, March JS. Research knowledge among the participants in the Treatment for Adolescents With Depression Study (TADS). J Am Acad Child Adolesc Psychiatry. 2007 Dec;46(12):1642-50. doi: 10.1097/chi.0b013e318153f8c7. PMID 18030086
- [Derived] May DE, Kratochvil CJ, Puumala SE, Silva SG, Rezac AJ, Hallin MJ, Reinecke MA, Vitiello B, Weller EB, Pathak S, Simons AD, March JS. A manual-based intervention to address clinical crises and retain patients in the Treatment of Adolescents With Depression Study (TADS). J Am Acad Child Adolesc Psychiatry. 2007 May;46(5):573-581. doi: 10.1097/chi.0b013e3180323342. PMID 17450048
- See also: NIMH Press Release — http://www.nimh.nih.gov/science-news/2007/depressed-adolescents-respond-best-to-combination-treatment.shtml